CLINICAL TRIAL: NCT02648425
Title: Phase I Study to Evaluate the Safety and Tolerability of ASLAN001 in Combination With Cisplatin and 5-Fluorouracil or Cisplatin and Capecitabine
Brief Title: Safety and Tolerability of ASLAN001 in Combination With Cisplatin and 5-FU or Cisplatin and Capecitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-002
Record Dates: First submitted 2015-06-21; First posted 2016-01-07 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumor
Keywords: ASLAN001; Varlitinib
MeSH Terms: interventions — ARRY-334543; Cisplatin; Capecitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A / Amended Regimen A (Experimental): Regimen A: Cisplatin + 5-fluorouracil
  ASLAN001 daily in combination with:
  Cisplatin 80 mg/m2 IV infusion for 1 day and 5-fluorouracil 800 mg/m2/day IV infusion for 5 days every 3 weeks for up to 6 cycles.
  Or
  Amended Regimen A: Cisplatin + 5-fluorouracil + leucovorin
  ASLAN001 daily in combination with:
  Cisplatin 35 mg/m2 24-hour infusion for day 1 and day 8, 5-fluorouracil 2,000 mg/m2 and Leucovorin 300mg/m2 24-hour infusion for day 1, day 8 and day 15 every 4 weeks for up to 6 cycles.
  Interventions: Drug: ASLAN001; Drug: cisplatin + 5-fluorouracil (or+ Leucovorin)
- Regimen B (Experimental): Regimen B: Cisplatin + capecitabine
  ASLAN001 daily in combination with:
  Cisplatin 60-80 mg/m2 IV infusion on Day 1 and capecitabine 1,000 mg/m2 orally BID for 14 days every 3 weeks for up to 6 cycles.
  Interventions: Drug: ASLAN001; Drug: cisplatin + capecitabine

INTERVENTIONS:
Drug: ASLAN001 — ASLAN001 400mg BID daily; ASLAN001 500mg BID daily; or ASLAN001 300mg BID daily
  Other Names: ARRY-334543; Varlitinib
Drug: cisplatin + capecitabine — Cisplatin 80 mg/m2 IV infusion and capecitabine 1,000 mg/m2 orally BID for 14 days every 3 weeks
  Arms: Regimen B
Drug: cisplatin + 5-fluorouracil (or+ Leucovorin) — Cisplatin 80 mg/m2 IV infusion and 5-fluorouracil 800 mg/m2/day IV infusion for 5 days every 3 weeks;
  Or
  Cisplatin 35 mg/m2 24-hour infusion for day 1 and day 8, 5-fluorouracil 2,000 mg/m2 and Leucovorin 300mg/m2 24-hour infusion for day 1, day 8 and day 15 every 4 weeks.
  Arms: Regimen A / Amended Regimen A

SUMMARY:
This is a phase IB study to assess the safety and tolerability of ASLAN001 when given in combination with either Cisplatin and 5-Fluorouracil or Cisplatin and Capecitabine, with a view to identifying the recommended Phase II dose.

DETAILED DESCRIPTION:
This is an open-label, Phase I, dose escalation study of ASLAN001 given in combination with Regimen A or Regimen B, in patients with metastatic solid tumors, eligible to receive the cisplatin/5-fluorouracil or cisplatin/capecitabine regimen.

Dose of ASLAN001 starts from 400mg BID; then, dose escalation to 500mg BID or dose de-escalation to 300mg BID will depend on DLTs observed in cohort.

Regimen A: Depends on preferred medical practice, Cohort 1A will receive ASLAN001 400 mg BID in combination with cisplatin 80 mg/m2 IV infusion and 5 fluorouracil 800 mg/m2/day IV infusion for 5 days every 3 weeks; or will receive ASLAN001 400 mg BID in combination with Cisplatin 35 mg/m2 24-hour infusion for day 1 and day 8, 5-fluorouracil 2,000 mg/m2 and Leucovorin 300mg/m2 24-hour infusion for day 1, day 8 and day 15 every 4 weeks.

Regimen B: Cohort 1B will receive ASLAN001 400 mg BID in combination with cisplatin 80 mg/m2 IV infusion and oral capecitabine 1,000 mg/m2 BID for 14 days every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 20 years of age or older at the time written informed consent is obtained.
2. Regimen A: Patients with metastatic solid tumors eligible for treatment with cisplatin and 5-fluorouracil. The standard dose and schedule of cisplatin and 5-fluorouracil will be according to the preference of investigators and institutions.

   Regimen B: Patients with metastatic solid tumors eligible for treatment with cisplatin in combination with capecitabine.
3. Patients with a partial gastrectomy may be allowed to participate in the study as long as they can take oral medications and meet all other inclusion/exclusion criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ and hematological function as evidenced by the following laboratory studies within 14 days prior to enrolment:

Hematological function, as follows:

* Absolute neutrophil count ≥ 1.5 x 109/L.
* Platelet count ≥ 100 x 109/L.
* Hemoglobin ≥ 9 g/dL.

Coagulation function, as follows:

* Partial thromboplastin time or activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN) per institutional laboratory normal range.
* International normalized ratio ≤ 1.5.

Renal function, as follows:

• Creatinine clearance ≥ 50 mL/min as calculated by Cockcroft-Gault formula.

Hepatic function, as follows:

* Total bilirubin ≤ 1.5 x ULN.
* AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present).

Exclusion Criteria:

1. Patients with persistent gastric outlet obstruction, complete dysphagia or feeding jejunostomy.
2. Patients receiving proton pump inhibitors or H2 antagonists for established, symptomatic gastro duodenal ulceration or gastroesophageal reflux disease.
3. Patients with unresolved toxicities of grade 2 or more from prior anti-cancer therapies.
4. Untreated or symptomatic central nervous system metastases. Patients with a history of brain metastases are eligible if definitive therapy has been administered (surgery and/or radiation therapy), there is no planned treatment for brain metastases, and the patient is clinically stable and is off corticosteroids for at least 2 weeks prior to enrolment.
5. Major surgical procedures within 28 days prior to enrolment.
6. Clinically significant cardiovascular diseases that are symptomatic or uncontrolled.
7. Known positive test for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen.
8. Pregnant or breast-feeding females.
9. Patients who have hearing impairment, due to the potential for ototoxicity of cisplatin.
10. Any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of ASALN001 | First 2 cycles
  Safety and tolerability as evaluated with:
  DLTs (in first 2 cycles); Maximum tolerated dose (MTD) of ASLAN001 in combination with cisplatin/capecitabine or cisplatin/5-FU will be determined.
Safety and Tolerability of ASALN001 | Baseline to post-dose
  Safety and tolerability as evaluated with:
  Adverse events.

SECONDARY OUTCOMES:
Preliminary assessment of the efficacy | Along the study duration
  •To provide a preliminary assessment of the efficacy of ASLAN001 when given in combination in Regimen A or Regimen B as measured by the objective response rate (ORR).
Pharmacokinetics profile (AUC) of ASLAN001 | Along the study duration
  To evaluate the pharmacokinetics of ASLAN001, when given in combination with Regimen A or Regimen B. Pharmacokinetic parameters including, but not limited to area under the plasma concentration-time curve (AUC) from 0 to 6 hours (AUC0-6).
Pharmacokinetics profile (Cmax) of ASLAN001 | Along the study duration
  To evaluate the pharmacokinetics of ASLAN001, when given in combination with Regimen A or Regimen B. Pharmacokinetic parameters including, but not limited to maximum plasma concentration (Cmax).
Pharmacokinetics profile (Cmin) of ASLAN001 | Along the study duration
  To evaluate the pharmacokinetics of ASLAN001, when given in combination with Regimen A or Regimen B. Pharmacokinetic parameters including, but not limited to minimum (trough) plasma concentration (Cmin).
Pharmacokinetics profile (RacAUC0-6) of ASLAN001 | Pharmacokinetic measurements will be from Cycle 1 Day 1 to Cycle 3 Day 1 (each cycle is 28 days for Amended Regimen A, and 21 days for Regimen A and B.
  To evaluate the pharmacokinetics of ASLAN001, when given in combination with Regimen A or Regimen B. Pharmacokinetic parameters including, but not limited to accumulation ratio for AUC (RacAUC0-6).
Pharmacokinetics profile (Tmax) of ASLAN001 | Along the study duration
  To evaluate the pharmacokinetics of ASLAN001, when given in combination with

CONTACTS AND LOCATIONS:
Overall Officials: ASLAN Pharma, Study Chair — ASLAN Pharmaceuticals
Locations (3):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei